CLINICAL TRIAL: NCT06914661
Title: Multicenter Real-world Study on the Efficacy and Safety of DS8201 in the Treatment of Metastatic Breast Cancer
Brief Title: Efficacy and Safety of DS8201 in Metastatic Breast Cancer's Treatment
Acronym: EASOFDIMBCT
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: DS8201
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Metastatic; Efficacy and Safety

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study analyzes the use of DS8201 in the treatment of metastatic breast cancer in the real world by analysis, exploring whether there are differences in effectiveness and safety between real-world conditions and clinical trials.

DETAILED DESCRIPTION:
In 2022, there were 19.96 million new cancer cases worldwide, of which about 2.3 million (11.6%) were new female breast cancer, making breast cancer the most common female malignant tumor. In China, 357.2 thousand new cases of female breast cancer were diagnosed, accounting for 15.6% of the total cases. Breast cancer ranks first in both morbidity and mortality among female tumors. About 3%-10% of newly diagnosed breast cancer patients have distant metastasis at the time of diagnosis, and about 30% of early breast cancer patients develop into advanced breast cancer. The 5-year survival rate of advanced breast cancer patients is only 20%, and the median overall survival time is 2-3 years. Breast cancer is mainly divided into four molecular subtypes, Luminal A, Luminal B, Human epidermal growth factor receptor2 (HER2) overexpression and triple-negative, with different treatment and prognosis. HER2 is important in breast cancer Driver genes AND outcome MEASURES. Because of the advent of HER2-targeting agents such as trastuzumab, guidelines classify HER2 as positive or negative. HER2 positivity (HER2+) was defined as HER2 IHC 3+, IHC 2+/ISH+ and represented 15% of the overall breast cancer population 20%, with a high degree of malignancy, strong invasion, poor prognosis, easy recurrence, easy metastasis. Her2-targeted drugs such as trastuzumab and pertuzumab have been clinically used to significantly prolong the survival of patients with HER2-positive breast cancer and improve the prognosis of the disease. With the advent of ADC drugs, patients with HER2 IHC1+ or IHC2+ and no HER2 amplification on in situ hybridization were defined as having low HER2 expression and occupying the breastAnd 45%-55% of patients with adenocarcinoma. Although these patients are not considered as an independent prognosis subtype at present, there are many new ADC drugs for treatment.

Novel antibody-drug conjugate (ADC). trastuzumab deruxtecan (hereafter, DS8201) is a combination of a HER2-targeting antibody and the DNA topoisomerase I inhibitor deruxtecan (DXd). DS8201 has the characteristics of loading new cytotoxic drugs, high drug-antibody ratio and high cell membrane permeability. Compared with traditional anti-HER2 drugs, DS8201 has anti-tumor effect on HER2 overexpression or low expression tumors NCT02564900 is an open-label, multicenter, first-in-human study phase I clinical trial to determine the safety and recommended dose of DS8201. The results of this study showed that the objective response rate was 59.5%(66/111) and the disease control rate was 93.7%(104/111) in 111 patients who could be evaluated. The recommended therapeutic dose of DS8201 was 5.4mg/kg, and the anti-tumor activity of DS8201 was also shown in patients with HER2-low advanced breast cancer. In terms of safety, the most common grade 3/4 adverse events were hematologic toxicities, including anemia (19/115,17%), neutropenia (16/115,14%), thrombocytopenia (9/115,8%), and leukopenia (10/115,9%). There are also gastrointestinal reactions. More prominently, the experiment reported interstitial lung disease or pneumonitis in 20 patients, two of which resulted in treatment-related deaths. Interstitial pneumonia comes into people's vision and becomes an important risk of DS8201. The efficacy and safety of the drug were further determined in a phase III trial. DS8201-A-U201 (DESTINY-Breast01, NCT03248492) was a phase 2, multicenter, open-enrollment trial investigating DS-8201 in previously treated subjects with HER2-positive, unresectable, and/or metastatic breast cancer. The results of this study showed that with DS-8201a (5.4 mg/kg), the ORR was 60.9% and the disease control rate (DCR) was 97.3% with a median follow-up time of 11.1 months. The median duration of response (DOR) was 14.8 months, and the median PFS was 16.4 months. This study showed that DS8201 showed reliable antitumor activity in patients with HER2-positive metastatic breast cancer who had failed multiple lines of therapy. In terms of safety, almost All patients (99.5%) who received the 5.4 mg/kg T-DXd dose had at least one adverse event; The incidence of adverse events of grade 3 or higher was 57%. The most common adverse event was neutropenia (20.7). Interstitial lung disease occurred in 13.6% of the patients and 4 of them died. DESTINY-Breast03 is a phase 3, multicenter, randomized, open-label, positively controlled trial evaluating DS-8201 as compared with T-DM1 in patients with HER2-positive, unresectable, and/or metastatic breast cancer previously treated with trastuzumab and a taxane. An exploratory analysis of PFS was performed for subsequent therapy after T-DXd treatment progression in this trial. The DESTINY-Breast03 trial compared the efficacy and toxicity of DS-8201 and trastuzumab emtancetuximab (T-DM1). The primary study median was progression-free survival (PFS), which was 28.8 months and 6.8 months, respectively. A 72% reduction in the risk of disease progression. In terms of safety, the incidence of adverse reactions of G3 or above in the two groups was 56% and 52%, respectively, and the incidence of interstitial pneumonia/pneumonitis was 15% and 3%, respectively, which cemented their status as second-line treatment. Since DESTINY-Breast03 excluded persons with clinically significant lung-specific disease, autoimmune disease, or connective-tissue and interstitial disease, the incidence of interstitial pneumonia was substantially lower than before. DESTINY-Breast04 is a phase III, multicenter, open-label, randomized, controlled trial evaluating DS-8201 versus physician's choice of treatment in patients with HER2-low, unresectable and/or metastatic breast cancer. These were defined as IHC 1+ and IHC 2+/ FISH-. The primary endpoint was PFS of 10.1 and 5.4 months in hormone receptor-positive patients, respectively. The incidence of G3 or worse adverse events was 52.6% and 67.4%, respectively. The incidence of interstitial pneumonia in T-Dxd group was 12.1%, and the frequency of death was 0.8%. The results suggest that T-DXd can consistently bring clinically significant improvements in PFS and OS compared with chemotherapy in patients with HER2-low metastatic breast cancer, regardless of HR status, and expand the population of T-Dxd from HER-2 positive to HER-2 low expression patients. Similar exclusion criteria for lung specific diseases were used in DESTINY-Breast04, and the incidence of interstitial pneumonia was controlled. The latest DB06 study released at the ASCO meeting in 2024 shows the successful exploration of DS8201 in the field of HER2 ultra-low expression, bringing new hope to breast cancer patients.

Based on its potent antitumor activity, T-DXd has been approved by the National Medical Products Administration for the treatment of adult patients with unresectable or metastatic HER2-positive breast cancer who have received at least one previous anti-HER2 drug therapy, and for the treatment of patients who have received at least one previous systemic therapy in the metastatic disease stage. Or adult patients with unresectable or metastatic HER2-low breast cancer that relapsed during or within 6 months after completion of adjuvant chemotherapy. Although TDXd has achieved remarkable efficacy in second-line and above advanced HER-2 positive breast cancer, there are often the following problems in the clinical application: (1) The recommended dose in our clinical trials is 5.4mg/kg, but in real life, due to the high cost of treatment, medical insurance funds can not cover and other economic factors, the actual clinical application of the most close to the full use of the whole dose, usually fail to reach the recommended dose (5.4mg/kg), there is insufficient dose. A real world study is needed to see if the current interventions have any impact on patient outcomes. (2) In the clinical trial, the enrolled patients were screened to a certain extent, and patients with clinically significant lung diseases were excluded, which reduced the incidence of adverse reactions of interstitial pneumonia. At the same time, the proportion of Asian population in clinical trials was often less than 50% (except DESTINY-Breast03, the proportion could reach 60% after adding the data from Korea and Japan). Based on this, it does not fully represent the actual efficacy in the Chinese population, and the consistency between the incidence of adverse reactions in the Chinese population and the clinical trial results needs to be explored in real world studies, especially the toxicity of interstitial pneumonia.

The aim of this study is to analyze the real-world clinical trial data to investigate the efficacy and safety of DS8201-containing formula in the treatment of HER2 positive and HER2 low expression advanced breast cancer patients in the real world, as well as the factors that may affect the efficacy, in order to provide some reference experience for the clinical application of DS8201.

ELIGIBILITY:
Inclusion criteria: (1) age ≥18 years old; (2) breast cancer confirmed by pathological diagnosis; (3) the presence of one or more distant metastatic lesions confirmed by pathology or imaging; (4) patients had received DS8201 treatment; (5) Complete medical records, complete blood routine and liver and kidney function test results during treatment.

Exclusion criteria: no history of traceable or missing clinical data.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
PFS | baseline and 1 year
  Time to disease progression or death from the first receipt of treatment in each line of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided